CLINICAL TRIAL: NCT00171561
Title: A 24-week Study to Evaluate the Effectiveness of Valsartan in Combination With Hydrochlorothiazide Versus Amlodipine on Arterial Compliance in Patients With Hypertension, Type 2 Diabetes and Albuminuria
Brief Title: Valsartan/Hydrochlorothiazide Combination vs Amlodipine in Patients With Hypertension, Diabetes, and Albuminuria.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631B2404
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: hypertension; diabetes; albuminuria; valsartan; hydrochlorothiazide; amlodipine
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Albuminuria | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: valsartan/hydrochlorothiazide

SUMMARY:
The purpose of this study is assess if treatment with valsartan and a diuretic, hydrochlorothiazide, has beneficial effects in people with high blood pressure, diabetes, and albuminuria (protein in the urine) compared with amlodipine. In particular, the study will assess whether the treatment will decrease the stiffness of the blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* elevated blood pressure and pulse pressure
* albuminuria

Exclusion Criteria:

* Severe hypertension
* History of stroke, myocardial infarction, heart failure, chest pain, abnormal heart rhythm
* Liver, kidney (not caused by diabetes), or pancreas disease
* Type 1 diabetes or uncontrolled type 2 diabetes
* Allergy to certain medications used to treat high blood pressure

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2003-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Blood measures of hypertension after 24 weeks

SECONDARY OUTCOMES:
Blood measures of hypertension in arterial system after 24 weeks
Change in protein excretion rate after 24 weeks
Change in serum markers of endothelial function and oxidative stress after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Karalliedde J, Maltese G, Hill B, Viberti G, Gnudi L. Effect of renin-angiotensin system blockade on soluble Klotho in patients with type 2 diabetes, systolic hypertension, and albuminuria. Clin J Am Soc Nephrol. 2013 Nov;8(11):1899-905. doi: 10.2215/CJN.02700313. Epub 2013 Aug 8. PMID 23929932